CLINICAL TRIAL: NCT03776396
Title: Perioperative Protocol Goal Directed Therapy in Kidney Transplantation: Fluid Therapy Optimization and Impact on Postoperative Complications.
Brief Title: Perioperative Goal Directed Therapy in Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Marinella Astuto, Principal Investigator, University of Catania
Other Study IDs: 31/2016/PO
Record Dates: First submitted 2018-12-06; First posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Kidney Transplant; Complications
Keywords: Perioperative Goal Directed Therapy; Minimally invasive hemodynamic monitoring; Kidney transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental cohort: 33 patient undergoing to kidney transplantation from cadaver at University Hospital "G. Rodolico" of Catania, in which an innovative Perioperative Goal Directed Therapy (PGDT) protocol will be used.
- Historical control group: 33 patients underwent to kidney transplantation from cadaver at University Hospital "G. Rodolico" of Catania in 2015, in which a PGDT protocol was not used, but a common hemodynamic monitoring, based on parameters such as central venous pressure and / or invasive arterial pressure, was performed.

SUMMARY:
In literature there is a huge amount of works demonstrating the direct correlation between volemic overload or fluid deficit and hypoperfusion and the increase in the rate of major postoperative complications in patients with high cardiovascular risk and chronic renal failure candidate to kidney transplantation from cadaver. It is also widely demonstrated that in certain populations with high surgical and post-operative complications risk, the adoption of targeted haemodynamic and clinical-therapeutic management protocols is indicated. The current trend is therefore to guarantee greater precision in the intraoperative management of patients undergoing kidney transplantation from cadaver by using a specific protocol that can be framed in the recent and innovative concept of Perioperative Gold Directed Therapy (PGDT), resulting from the adoption of an advanced minimally invasive hemodynamic monitoring technology with a special sensor called FloTrac (Edwards Lifesciences), already extensively tested in an extensive case series of high perioperative risk patients underwent to major abdominal surgery, major vascular surgery, major orthopedic surgery and cardio-thoracic surgery. In the present study there will be enrolled all patients who are candidates for kidney transplant from cadaver at the University Hospital "G. Rodolico" of Catania that meet the inclusion criteria of the study and will give their informed consent to participation. The enrolled patients will be monitored for a maximum period of 7 days from transplantation. As control group there will be considered an historical cohort of patients who underwent kidney transplantation from cadaver in 2015, in which a PGDT protocol was not used, but a common hemodynamic monitoring, based on parameters such as central venous pressure and / or invasive arterial pressure, was performed according to the international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Classification III-IV;
* Age between 18 and 65 years;
* First kidney transplantation from cadaver;
* Absence of atrial fibrillation or severe arrhythmia;
* Informed consent.

Exclusion Criteria:

* Lack of informed consent;
* Age less that 18 or greater than 65 years;
* Atrial fibrillation and high frequency tachyarrhythmias;
* Previous transplantation from cadaver.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 33 consecutive patients candidates for kidney transplantation from cadaver that meet the eligibility criteria of the study and 33 patients who underwent kidney transplantation in 2015
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Frequency rate of postoperative complications | 7 days after transplantation
  The frequency rate of the subsequent postoperative complications in the two study cohort will be determined: early postoperative pulmonary complications (prolonged mechanical ventilation, failure acute respiratory disease, acute pulmonary edema, pulmonary infections); major cardiovascular complications (ischemic cardiac events and heart failure congestive); major surgical complications (anastomosis, delayed postoperative ileum, nausea and postoperative vomiting).
Duration of hospitalization in a semi-intensive and intensive hospital ward. | 7 days after transplantation

SECONDARY OUTCOMES:
Number of patients with delayed graft failure in the two study cohorts | 7 days after transplantation
Number of patients requiring hemodialysis in the two study cohorts | 7 days after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- "G. Rodolico" Presidium of the Azienda Ospedaliero Universitaria "Policlinico-Vittorio Emanuele", Catania, Italy